CLINICAL TRIAL: NCT03787745
Title: The Effect of Ischemic Postconditioning in Patients With STEMI Undergoing Primary PCI (DANAMI4-iPOST2)
Brief Title: Ischemic Postconditioning in STEMI Patients Treated With Primary PCI
Acronym: iPOST2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Thomas Engstrom, Professor, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-18051256
Record Dates: First submitted 2018-12-19; First posted 2018-12-26 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: ST Segment Elevation Myocardial Infarction
Keywords: Primary PCI; Ischemic postconditioning; Clinical outcome
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Ischemic Postconditioning; Congresses as Topic

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, placebo controlled
Who Masked: Outcomes Assessor
Masking Description: All study personell involved in outcome assessment will be blinded to the treatment employed
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ischemic postconditioning (Active Comparator): In addition to state of the art primary PCI in patients with TIMI0-1 ischemic postconditioning with an adequately sized balloon (60 reperfusion/60 seconds re-occlusion, four cycles) will be performed, however thrombectomy will not be allowed
  Interventions: Procedure: Ischemic postconditioning
- Conventional (Placebo Comparator): State of the art primary PCI in patients with TIMI0-1 will be performed, however thrombectomy will not be allowed
  Interventions: Procedure: Conventional

INTERVENTIONS:
Procedure: Ischemic postconditioning — After 60 seconds of reperfusion, ischemic postconditioning with an adequately sized balloon (60 reperfusion/60 seconds re-occlusion, four cycles) will be performed
  Arms: Ischemic postconditioning
Procedure: Conventional — State of the art primary PCI, however thrombectomy is not allowed
  Arms: Conventional

SUMMARY:
In a prospective, randomized clinical trial the iPOST2 trial will determine whether ischemic postconditioning reduces reperfusion injury and this will translate into improved clinical outcome of heart failure and death for STEMI patients who present with TIMI0-1 undergoing primary PCI

DETAILED DESCRIPTION:
Myocardial reperfusion with the use primary percutaneous coronary intervention (PCI) is effective, but restoration of blood flow may itself jeopardize the myocardium, a phenomenon known as reperfusion injury.

In ischemic postconditioning (iPOST), repetitive interruptions of blood flow to the injured region applied after initial reperfusion, has been shown favorable with different modalities such as biomarkers, echocardiography and cardiac magnetic resonance.

However, the largest trial to date (DANAMI3-iPOST) failed to show clinical favor of iPOST when compared to conventional PCI. Importantly, however, in DANAMI3-iPOST thrombectomy was allowed and this might have impaired postconditioning, since thrombectomy itself creates reperfusion and thus reperfusion damage. Analysis of the fraction of DANAMI3-iPOST patients not undergoing thrombectomy showed a remarkable 45% reduction in death and heart failure in favor of postconditioning.

iPOST2 will investigate in a randomized, prospective and adequately powered trial the effect of iPOST without thrombectomy compared to conventional PCI on the development of heart failure and death in STEMI patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Acute onset of chest pain with < 12 hours duration
* STEMI as characterized by 2 mm ST elevation in 2 or more V1 through V4 leads or presumed new left bundle branch block with minimum of 1 mm concordant ST elevation or 1 mV ST-segment elevation in the limb lead (II, III and aVF, I, aVL) and V4-V6 or ST depression in 2 or more V1 through V4 leads indicating posterior AMI.
* TIMI flow 0-1 in infarct related artery

Exclusion Criteria:

* Potential pregnancy
* Refusal to participate
* OHCA without subsequent consciousness despite ROSC
* Thrombectomy considered unavoidable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1800 (Estimated)
Dates: Start 2019-02-04 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2033-01-31 (Estimated)

PRIMARY OUTCOMES:
All cause mortality or hospitalization for heart failure | From date of randomization until the date of first documented hospitalization for heart failure or date of death from any cause, whichever came first, assessed up to 280 events have been adjudicated or up to 36 months
  Composite endpoint of all cause mortality or hospitalization for heart failure which ever occur first

SECONDARY OUTCOMES:
All cause mortality | From date of randomization until the date of first documented death from any cause assessed up to 280 events have been adjudicated or up to 36 months
  All cause mortality
Percentage of patients hospitalized for heart failure | From date of randomization until the date of first documented hospitalization for heart failure assessed up to 280 events have been adjudicated or up to 36 months
  Any hospitalization for heart failure occurring after the index STEMI
Percentage of patients with myocardial infarction | From date of randomization until the date of first documented hospitalization for heart failure or date of death from any cause, whichever came first, assessed up to 280 events have been adjudicated or up to 36 months
  Any myocardial infarction occurring after the index STEMI
Cardiovascular death | From date of randomization until the date of first documented hospitalization for heart failure or date of death from any cause, whichever came first, assessed up to 280 events have been adjudicated or up to 36 months
  Cardiovascular death
Percentage of patients with stroke | From date of randomization until the date of first documented hospitalization for heart failure or date of death from any cause, whichever came first, assessed up to 280 events have been adjudicated or up to 36 months
  An acute episode of focal or global neurological dysfunction caused by brain injury
Percentage of patients with a combination of all-cause mortality, hospitalization for heart failure, new myocardial infarction and stroke/transitory cerebral ischemia | From date of randomization until the date of first documented hospitalization for heart failure or date of death from any cause, whichever came first, assessed up to 280 events have been adjudicated or up to 36 months
  Composite endpoint of all-cause mortality, hospitalization for heart failure, new myocardial infarction and stroke/transitory cerebral ischemia
Percentage of patients with a combination of hospitalization for heart failure and cardiovascular death | From date of randomization until the date of first documented hospitalization for heart failure or date of death from any cause, whichever came first, assessed up to 280 events have been adjudicated or up to 36 months
  A composite of hospitalization for heart failure and cardiovascular death
Danish eq5d5l standard Quality of life | 1 year
  Self assesed quality of life after the Danish eq5d5l standard scale (1 worst score -100 best score)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Engstrøm, DMSci, Study Chair — Rigshospitalet, Denmark
Locations (1):
- The Heart Center, Rigshospitalet, University of Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Engstrom T, Kelbaek H, Helqvist S, Hofsten DE, Klovgaard L, Clemmensen P, Holmvang L, Jorgensen E, Pedersen F, Saunamaki K, Ravkilde J, Tilsted HH, Villadsen A, Aaroe J, Jensen SE, Raungaard B, Botker HE, Terkelsen CJ, Maeng M, Kaltoft A, Krusell LR, Jensen LO, Veien KT, Kofoed KF, Torp-Pedersen C, Kyhl K, Nepper-Christensen L, Treiman M, Vejlstrup N, Ahtarovski K, Lonborg J, Kober L; Third Danish Study of Optimal Acute Treatment of Patients With ST Elevation Myocardial Infarction-Ischemic Postconditioning (DANAMI-3-iPOST) Investigators. Effect of Ischemic Postconditioning During Primary Percutaneous Coronary Intervention for Patients With ST-Segment Elevation Myocardial Infarction: A Randomized Clinical Trial. JAMA Cardiol. 2017 May 1;2(5):490-497. doi: 10.1001/jamacardio.2017.0022. PMID 28249094